CLINICAL TRIAL: NCT03138551
Title: Examining Relationships Between Family Mealtime Routines and Feeding Outcomes in Young Children With Sensory Food Aversions
Brief Title: Examining Relationships Between Family Mealtime and Feeding Outcomes in Young Children With Sensory Food Aversions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Angela Caldwell, Assistant Professor, University of Pittsburgh
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO15060533
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Feeding Disorder of Infancy or Early Childhood
Keywords: Sensory Food Aversions

STUDY DESIGN:
Intervention Model Description: Single-Case Experimental Design
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mealtime PREP (Experimental): Every participant enrolled in this single-case experimental design trial with multiple replications progressed through three phases.
  A: Baseline - typical mealtimes in the home.
  B: Parent-Training - parents trained in Mealtime PREP (Promoting Routines of Exploration and Play) intervention.
  B-prime: Family Autonomy - parents continue to deliver treatment strategies. Therapist support withdrawn.
  Interventions: Behavioral: Mealtime PREP (Promoting Routines of Exploration and Play)

INTERVENTIONS:
Behavioral: Mealtime PREP (Promoting Routines of Exploration and Play)

SUMMARY:
This study will examine the feasibility and preliminary effects of the Mealtime PREP (Promoting Routines of Exploration and Play) intervention package for young children with Sensory Food Aversions and their parents.

DETAILED DESCRIPTION:
This pilot study will collect rich data from twenty participants on the feasibility and effects of a novel intervention, the Mealtime PREP, which has a dyadic focus on both the young child and the parent participants. The investigators will collect video recorded child meals in the home during a baseline period (under normal circumstances), during parent-training (while parents are practicing skills learned), and following parent training (when therapist support is withdrawn). This in depth examination of child meals will provide valuable information to guide the optimization of this intervention approach for future trials.

ELIGIBILITY:
Inclusion Criteria:

* Child must meet all criteria of the diagnosis of Sensory Food Aversions

  1. The child consistently refuses to eat specific foods with specific tastes/textures and/or smells.
  2. Onset of food refusal occurs during the introduction of a novel type of food (e.g., the child may drink one type of milk but refuse another, may eat carrots but refuse green beans, may drink milk but refuse baby food).
  3. The child eats without difficulty when offered preferred foods.
  4. The food refusal causes specific nutritional deficiencies or delay of oral motor development.
* Parent is able to read, write, speak and understand English.

Exclusion Criteria: None

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-10-11 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Food Acceptance | 30 meals video recorded throughout study participation (10 per phase, 1 month)
  Significant change in percentage of targeted food accepted between phases.

SECONDARY OUTCOMES:
3-Day Food Diary | Baseline through Study Completion (1 month)
  Increased number of foods eaten over a three-day period.
Behavioral Pediatric Feeding Assessment (BPFAS) | Baseline through Study Completion (1 month)
  Clinically relevant change in child feeding behavior and/or parental report of mealtime problems.

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Caldwell, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Caldwell AR, Skidmore ER, Raina KD, Rogers JC, Terhorst L, Danford CA, Bendixen RM. Behavioral Activation Approach to Parent Training: Feasibility of Promoting Routines of Exploration and Play During Mealtime (Mealtime PREP). Am J Occup Ther. 2018 Nov/Dec;72(6):7206205030p1-7206205030p8. doi: 10.5014/ajot.2018.028365. PMID 30760395